CLINICAL TRIAL: NCT02363062
Title: Identification of New Genes Causing Frontotemporal Lobar Degeneration by Whole Exome Sequencing and Characterization of the Associated Phenotypes
Brief Title: Identification of New FTLD Genes
Acronym: FTLD-Exome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A00157-40
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2016-08

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: frontotemporal lobar degeneration; genes; whole exome sequencing
MeSH Terms: conditions — Frontotemporal Lobar Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be collected by a nurse, during a single consultation or hospitalization
Oversight: Data Monitoring Committee: No

SUMMARY:
The major objective of the project is to map/identify new loci/genes, by a combination of whole exome sequencing and genome-wide linkage in autosomal dominant FTLD families excluded for known mutations.

Several secondary goals will be attained in the course of during the project:

For each novel gene identified in this project, we will determine the spectrum of mutations, evaluate their frequency and characterize the associated phenotypes. This will allow us to establish genotype-phenotype correlations in a large number of families, which will improve the nosology of these disorders and the diagnostic procedures;

DETAILED DESCRIPTION:
Background and justification of the research. In France, 6,000 to 8,000 patients are affected by frontotemporal lobar degeneration (FTLD). FTLD are degenerative dementias related to Alzheimer's disease, characterized by behavioural, language and cognitive disorders beginning in the sixth decade. The genetic forms of FTLD are frequent (30-50% of the patients), but the genes responsible for 30-40% of familial FTLD are still unknown. At present, no molecular diagnosis can be proposed for 30% of the FTLD families and patients, for which the responsible genes are still unknown. No presymptomatic testing can be proposed either to at-risk relatives in these families.

Objectives.

1. The principal objective of this proposal is to identify one or several genes responsible for FTLD.
2. The secondary objectives are to:

   * evaluate the relative frequency of identified genes;
   * describe the phenotypes associated with the mutations in these genes;
   * establish phenotype-genotype correlations in order to improve the diagnostic procedures and strategies;
   * develop new genetic diagnostic analyses in the near future.

Project The patients will be recruited in three hospitals (Paris Salpetriere, Limoges, Lille). These three centers are partners of a national clinico-genetic network of 20 french centers experts in FTLD/FTLD-ALS, coordinated by Dr. I Le Ber. The participants in this network have collaborated for the last 15 years, and have already recruited over 1,000 patients with FTLD. Sequencing of known genes in these families allowed the identification of 150 families with an autosomal dominant form of FTLD not associated with a known mutation. Through the network, we aim to recruit 400 new patients with FTLD during the 4 years of the project. This estimation is based on the annual recruitment of the network during the last two years.

In this project, the 30 most informative families will be extended (440 patients and relatives sampled).

The combination of whole exome sequencing with genetic linkage studies in FTLD families without known mutations, and the large number of families included in this project, are two major points that should lead to the identification of several new genes. When causative genes are identified, we will establish the frequencies of mutations, extend the mutational spectrum, describe the clinical phenotypes and establish phenotype-genotype correlations. Genetic parameters such as penetrance will be analyzed.

ELIGIBILITY:
Patients are included if they:

i) are affected by FTLD±ALS according to the international diagnosis criteria and ii) Have (or their legal representatives have) given signed written informed consent for the research.

iii) are affiliated to social security or beneficiary of such régime

Relatives are included if they:

i) are aged >18 years and ii) Have signed an informed consent for the research. are affiliated to social security or beneficiary of such

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by FTLD±ALS according to the international diagnosis criteria and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2015-02-02 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
whole exome sequencing | Day 1
  genes responsible for FTLD /Blood samples will be collected by a nurse, during a single consultation or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LE BER, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitié Salpetriere Hospital, Paris, France

REFERENCES:
- [Derived] Ceslis A, Argall R, Henderson RD, McCombe PA, Robinson GA. The spectrum of language impairments in amyotrophic lateral sclerosis. Cortex. 2020 Nov;132:349-360. doi: 10.1016/j.cortex.2020.09.003. Epub 2020 Sep 18. PMID 33031977
- [Derived] Didic M, Aglieri V, Tramoni-Negre E, Ronat L, Le Ber I, Ceccaldi M, Belin P, Felician O. Progressive phonagnosia in a telephone operator carrying a C9orf72 expansion. Cortex. 2020 Nov;132:92-98. doi: 10.1016/j.cortex.2020.05.022. Epub 2020 Aug 10. PMID 32961393